CLINICAL TRIAL: NCT07288476
Title: Shareholder-driven Co-design and Piloting of Spanish Educational Videos About High Yield Pediatric Oncology Topics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-0595.cc; NCI-2025-08026 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2025-01-22; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cancer
Keywords: Spanish Speaking
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot educational videos (Experimental): Pilot education videos with Spanish-speaking parents as a tool to improve caregiver knowledge, satisfaction, confidence in caring for their child, and level of overwhelm.
  Interventions: Other: educational video

INTERVENTIONS:
Other: educational video — Spanish-language video to impart knowledge and understanding to parents caring for children with cancer

SUMMARY:
Families of children with cancer who speak languages other than English experience inequalities in healthcare, but little research has been done on solutions to improve care for these families. This study will partner parents with medical interpreters and clinicians to create educational videos about key cancer topics in Spanish and test their use as a tool to improve caregiver knowledge and experience in the setting of a language barrier. The project will lead to a future career development award application that increases the number of available languages and studies how multilingual educational videos impact caregiver knowledge and experience

ELIGIBILITY:
Inclusion Criteria:

Aims 1 and 2 (Video Development Phase):

* Legal caregiver aged ≥18 years of a child/young adult (0-25 years) undergoing active cancer treatment in low-intensity phases or off therapy.
* Native or fluent Spanish speaker.
* Willing and able to provide verbal consent.
* Willing to comply with study procedures and be available for the study duration.

Aim 3 (Video Pilot Phase):

* Legal caregiver aged ≥18 years of a child/young adult (0-25 years) with newly diagnosed or relapsed/refractory cancer (≤1 month).N
* Native or fluent Spanish speaker.
* Requires an interpreter for medical conversations.
* Willing and able to provide verbal consent.
* Willing to comply with study procedures and be available for the study duration.

Exclusion Criteria:

Aims 1 and 2:

* Insufficient cognitive functioning to complete study procedures (as determined by PI).
* Caregiver of a child/young adult who did not receive cancer-directed therapy.
* Caregiver of a child/young adult receiving high-intensity cancer treatment.
* Unable to read and speak Spanish fluently.

Aim 3:

* Insufficient cognitive functioning to complete study measures (as determined by PI).Caregiver of a child/young adult who did not receive cancer-directed therapy.
* Caregiver of a child/young adult not receiving cancer-directed therapy.
* Diagnosis of new or relapsed/refractory cancer occurred >1 month prior to enrollment.
* Unable to speak Spanish fluently.
* Does not require an interpreter for medical conversations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Implementing a Spanish-Language Educational Video Intervention | 6 months
  The feasibility of implementing a Spanish-language educational video intervention will be assessed using the Feasibility of Intervention measure.
Acceptability of Implementing a Spanish-Language Educational Video Intervention | 6 months
  The acceptability of the Spanish-language educational video intervention will be assessed using the Acceptability of Intervention Measure.

SECONDARY OUTCOMES:
Impact on caregiver knowledge measured by post-intervention surveys | 12 months
  The impact of the intervention on caregivers knowledge will be assessed through post-intervention questionnaires measuring changes in knowledge about caregiving, satisfaction with the educational material, and confidence in caring for their child.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided